CLINICAL TRIAL: NCT00079794
Title: Iscar for Supplemental Care in Stage IV Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001020-01 (NIH); Rosenzweig
Record Dates: First submitted 2004-03-15; First posted 2004-03-16 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Lung Cancer
Keywords: lung cancer; herbal medicine; non-small cell cancer; Iscar; mistletoe
MeSH Terms: conditions — Lung Neoplasms

INTERVENTIONS:
Drug: Iscar
Drug: mistletoe

SUMMARY:
The purpose of this study it to determine whether supplemental treatment with Iscar improves immune function and quality of life among Stage IV non-small cell lung carcinoma patients receiving conventional chemotherapy. Iscar is an herbal medicine made from the total plant extract of mistletoe. this preparation is already in use in Europe and its use in the US is likely to increase as cancer patients continue to seek alternative therapies.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Stage IV NSCLC patients who receive standard chemotherapy

Exclusion criteria:

* Known allergy to Viscum Album L.
* Concomitant use of other mistletoe products
* Concomitant use of mushroom glucan and proteoglycan extracts
* Concomitant use of thymus extract products
* Inability to self-report quality of life utilizing assessment tools
* Ongoing steroid or ACTH therapy
* Co-morbid immunocompromised state
* Pregnancy
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2001-09; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenzweig, MD, Principal Investigator — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States